CLINICAL TRIAL: NCT00996398
Title: Cold Water Immersion Does Not Reduce Knee Joint Position Sense in Healthy Participants: a Randomised Cross-over Trial'
Brief Title: Cold Water Immersion Does Not Reduce Knee Joint Position Sense in Healthy Participants: a Randomised Cross-over Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Dr. Alan Donnelly, University of LImerick
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ULREC 09/11
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Knee Joint Position Sense
Keywords: Cryotherapy; Joint Position Sense; Proprioception; Pre Cooling; Knee Injury; Physical Therapy Modalities; Physical Therapy Techniques; Weightbearing; NonWeightbearing; Randomised Control Trial
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cold water immersion (Experimental): 14°C ± 1°C for the cold water immersion for 30 minutes to the level of the umbilicus
  Interventions: Other: Tepid water immersion

INTERVENTIONS:
Other: Tepid water immersion — 28°C ± 1°C for the cold water immersion for 30 minutes to the level of the umbilicus

SUMMARY:
The aim of this project is to assess the effect of cold water immersion on knee joint re-positional sense in healthy subjects. Cryotherapy, in the form of cold water immersion, had previously been shown to improve athletic performance however, debate exists within the existing literature regarding whether proprioception, in the form or joint position sense, is effected post treatment.

Null hypothesis (H0): Water immersion has no effect on joint position sense (JPS).

Alternate hypothesis (H1): Water immersion has an effect on joint position sense.

DETAILED DESCRIPTION:
This was a prospective, randomised, cross-over design where volunteers acted as their own controls. The volunteers were immersed at two temperatures (detailed below) and these sessions were separated by six to ten days. The order of the testing was randomly assigned using a random number generator. Ethical approval of the design of this trial was gained from the University of Limerick's Research Ethics Committee and signed informed consent was gained from each participant before any data collection took place.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of 18 and 40 who complete both a Par-Q test and sign an informed consent form.

Exclusion Criteria:

* Potential subjects who do not complete a Par-Q questionnaire or provide written consent. Subjects with any ankle or knee injuries in the past twelve months.
* Students who have a recent history of ear or vestibular conditions.
* Subjects who will not be available to attend all sessions.
* Subjects who are under the age of 18 or over the age of 40.
* Subjects who aren't comfortable with being blind-folded or videotaped during testing.
* Those who are sensitive to cold exposure or show signs of a contraindication to cryotherapy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Knee Joint Position Sense | 10 minutes pre and 5 minutes post immersion

CONTACTS AND LOCATIONS:
Overall Officials: Alan E Donnelly, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Limerick, Ireland